CLINICAL TRIAL: NCT04574011
Title: Prediction of Fluid Responsiveness With Non-invasive Dynamic Parameters in Spontaneous Breathing Patients
Brief Title: Fluid Responsiveness in Spontaneously Ventilating Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: H-2010-013-1161
Record Dates: First submitted 2020-09-23; First posted 2020-10-05 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Fluid Responsiveness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluid challenge responder (Experimental): If the ratio of the stroke volume change after passive leg raising is the same or larger than 10%, the patient is assigned to RESPONDER group.
  Interventions: Diagnostic Test: Passive leg raising
- Fluid challenge non-responder (Experimental): If the ratio of the stroke volume change after passive leg raising is less than 10%, the patient is assigned to RESPONDER group.
  Interventions: Diagnostic Test: Passive leg raising

INTERVENTIONS:
Diagnostic Test: Passive leg raising — Raise the patient's lower limb at a 45 degree angle while lying down

SUMMARY:
The purpose of this study is to find out if non-invasive dynamic parameters can predict fluid responsiveness in spontaneous breathing patients.

DETAILED DESCRIPTION:
Knowing when to give fluids to the patient is very important in fluid therapy.It is appropriate to administer it to patients whose cardiac output will increase when the fluid is administered (a patient with fluid responsiveness). Appropriate fluid administration can hemodynamically stabilize the patient's condition and reduce unnecessary fluid administration, thereby reducing complications that occur when fluid is insufficient or excessive fluid is administered.

The most commonly used dynamic variables in clinical practice are pulse pressure variation (PPV), stroke volume variation (SVV), and systolic pressure variation that can be obtained by invasive arterial tube insertion. However, recently a non-invasive monitoring method is being used in more and more areas, and in many cases it is necessary to closely monitor the patient's hemodynamic status without mounting an arterial catheter. Therefore, if the variables measured by a non-invasive method can predict fluid responsiveness at a reliable level, it will be of great help in clinical practice.

According to previous studies, dynamic variables can relatively accurately predict fluid responsiveness only in patients undergoing mechanical ventilation. However, in actual clinic, it is necessary to evaluate fluid reactivity even in patients who are not under mechanical positive pressure ventilation. Accurate fluid treatment should be performed during or after surgery under spinal anesthesia in the recovery room. In addition, there are cases in which dynamic variables must be monitored non-invasively in spontaneous breathing patients who do not undergo mechanical ventilation even in intensive care units.

It is clinically meaningful to predict fluid responsiveness in spontaneous breathing patients using such a non-invasive method of monitoring. However, there is limited data on how to evaluate fluid responsiveness in these patient groups. Therefore, the purpose of this study is to evaluate whether fluid responsiveness can be predicted in spontaneous breathing patients using non-invasive dynamic variables.

ELIGIBILITY:
Inclusion Criteria:

* for patients undergoing surgery under actual spinal anesthesia whose estimated blood loss during surgery is moderate to high (e.g. total knee arthroplasty, total hip arthroplasty)
* Patients with a history of cerebrovascular disease
* Patients with a history of 1 or 2 vessel disease
* Left ventricle ejection fraction (LVEF) Patients with 30% or more and less than 55% of these patients
* Patients who need close hemodynamic monitoring during operation
* ASA (American Society of Anesthesiology) physical status classification system I, II, III
* no difficulty in passive leg raising maneuver

Exclusion Criteria:

* Patients unable to communicate
* Patients who cannot or have difficulty in PLR (passive leg raising) maneuver (patients who cause pain when performing PLR due to trauma of the lower extremities, patients with spine disease that causes pain during PLR, and patient applying splint due to a fracture of the lower extremity)
* Patients unable to attach the finger cuff of the ClearSight sytem to one of the fingers of both hands. (Patients applying a splint due to a fracture of both upper limbs, etc.)
* Patients unable to perform transthoracic ultrasound examination (multiple trauma patients with rib fracture, etc.)
* Patients having difficulty obtaining blood pressure waveforms through the ClearSight system due to poor peripheral vascular perfusion (uncontrolled diabetes patients, patients with peripheral vascular disease, etc.)
* Patients with arrhythmia with moderate or higher risk such as atrial fibrillation or atrial flutter
* Heart failure patients with less than 30% of the left ventricular ejection fraction(LVEF) on echocardiography or patients with moderate to severe left ventricular wall motor dysfunction, or patients with cardiovascular disease of 3 vessel disease
* Other patients who are not appropriate to participate in the study as judged by the researcher

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-03-05 (Estimated); Primary Completion 2021-06-11 (Estimated); Study Completion 2021-07-21 (Estimated)

PRIMARY OUTCOMES:
ClearSight PPV | before induction, 20 minutes
  Pulse pressure variation measured by ClearSight System arterial waveform

SECONDARY OUTCOMES:
ClearSight SVV | before induction, 20 minutes
  Stroke volume variation measured by ClearSight System
normal ventilation △IVC (inferior vena cava) diameter | before induction, 20 minutes
  △IVC diameter variation on normal ventilation
augmented ventilation △IVC (inferior vena cava) diameter | before induction, 20 minutes
  △IVC diameter variation on augmented ventilation
normal ventilation △POP (pulse oximeter plethysmography) | before induction, 20 minutes
  △POP on normal ventilation
augmented ventilation △POP (pulse oximeter plethysmography) | before induction, 20 minutes
  △POP on augmented ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Jintae Kim, M.D, Principal Investigator — SNUH
Locations (1):
- Seoul National University Hospital, Seoul, Jongro-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cavallaro F, Sandroni C, Antonelli M. Functional hemodynamic monitoring and dynamic indices of fluid responsiveness. Minerva Anestesiol. 2008 Apr;74(4):123-35. Epub 2008 Jan 24. PMID 18212731
- [Background] Drvar Z, Pavlek M, Drvar V, Tomasevic B, Baronica R, Peric M. [Stroke volume and pulse pressure variation are good predictors of fluid responsiveness in sepsis patients]. Acta Med Croatica. 2013 Dec;67(5):407-14. Croatian. PMID 24979881
- [Background] Cecconi M, Monge Garcia MI, Gracia Romero M, Mellinghoff J, Caliandro F, Grounds RM, Rhodes A. The use of pulse pressure variation and stroke volume variation in spontaneously breathing patients to assess dynamic arterial elastance and to predict arterial pressure response to fluid administration. Anesth Analg. 2015 Jan;120(1):76-84. doi: 10.1213/ANE.0000000000000442. PMID 25230102
- [Background] Slagt C, Malagon I, Groeneveld AB. Systematic review of uncalibrated arterial pressure waveform analysis to determine cardiac output and stroke volume variation. Br J Anaesth. 2014 Apr;112(4):626-37. doi: 10.1093/bja/aet429. Epub 2014 Jan 14. PMID 24431387
- [Background] Vos JJ, Poterman M, Salm PP, Van Amsterdam K, Struys MM, Scheeren TW, Kalmar AF. Noninvasive pulse pressure variation and stroke volume variation to predict fluid responsiveness at multiple thresholds: a prospective observational study. Can J Anaesth. 2015 Nov;62(11):1153-60. doi: 10.1007/s12630-015-0464-2. Epub 2015 Sep 3. PMID 26335905
- [Background] Thiel SW, Kollef MH, Isakow W. Non-invasive stroke volume measurement and passive leg raising predict volume responsiveness in medical ICU patients: an observational cohort study. Crit Care. 2009;13(4):R111. doi: 10.1186/cc7955. Epub 2009 Jul 8. PMID 19586543
- [Background] Chaves RCF, Correa TD, Neto AS, Bravim BA, Cordioli RL, Moreira FT, Timenetsky KT, de Assuncao MSC. Assessment of fluid responsiveness in spontaneously breathing patients: a systematic review of literature. Ann Intensive Care. 2018 Feb 9;8(1):21. doi: 10.1186/s13613-018-0365-y. PMID 29427013